CLINICAL TRIAL: NCT06282887
Title: The Effects of Music Therapy on Improving Psychological States of Cancer Patients Undergoing MRI Scans and a Relevant Mediator
Brief Title: Effects of Music Therapy on Psychological States Among Cancer Patients Undergoing MRI Scans and a Relevant Mediator
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Guangzhou Concord Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 2021-IIT-002
Record Dates: First submitted 2023-11-05; First posted 2024-02-28 (Actual); Last update posted 2025-01-01 (Actual); Status verified 2024-11

CONDITIONS: Psycho-Oncology
Keywords: MRI; Anxiety; Symptom distress; Relaxation; Music therapy
MeSH Terms: conditions — Anxiety Disorders | interventions — Music Therapy

STUDY DESIGN:
Who Masked: Participant, Care Provider
Masking Description: All participants will be wearing a headphone, and they will not know if there will be music until they experience and finish the scan process.
  Radiographers are blinding to avoid biases.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Music Therapy Group (Experimental): Participants in the Music Therapy Group will receive standard care and approximately 15 minutes of music therapy before the MRI scan and will have music played through their headphones during the scanning process.
  Interventions: Other: Music therapy
- Control Group (No Intervention): Participants in the Control Group will receive standard care throughout the awaiting period and the scanning process.

INTERVENTIONS:
Other: Music therapy — The intervention has two parts. The first part is an approximately 15-minute music therapy session to induce relaxation and positive memories attached to the relaxing live music provided by a credentialed music therapist. The second part is music listening during the scanning process.
  Arms: Music Therapy Group

SUMMARY:
The primary objective of this study is to examine the effects of a music therapy protocol on improving anxiety, symptom distress, and relaxation among cancer patients who are going through MRI scanning. Physiological data, such as pulse rates and respiration rates will be collected. Furthermore, data about scanning efficiency will be collected to assess if scanning efficiency is affected by the protocol implementation. The secondary study objective is to assess whether or not there is a relationship between patient attention to music during the intervention process and the changes in anxiety, symptom distress, and relaxation.

DETAILED DESCRIPTION:
To assess the protocol, recruited participants will be randomly allocated into two groups: a control group or a music therapy group. Participants in the control group will receive standard care as usual, and they will be offered music therapy interventions upon their request during subsequent appointments. Participants in the music group will receive standard care and music therapy interventions. All participants will rate their psychological states pre- and post-MRI exams. Their physiological data will be recorded during the examination. After the scanning, they will complete an experience review.

ELIGIBILITY:
Inclusion Criteria:

1. The subject is diagnosed with cancer;
2. The subject is between 18- 60 years old;
3. The subject understands Mandarin, Cantonese, or English;
4. The subject did not use medication for sedatives, anxiolytics, and/or sleep aids;
5. The subject is awake without cognitive disorders;
6. the subject rates more than 0 on the 0-10 VAS for anxiety;
7. The subject has finished primary school level education.

Exclusion Criteria:

1. The subject withdraws the MRI scan;
2. The subject needs other intervention(s) to complete the scan;
3. The subject has hearing and/or visual impairments;
4. The subject has a history of a severe somatic psychiatric disease or clinically diagnosed mental disorders.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 80 (Estimated)
Dates: Start 2021-11-09 (Actual); Primary Completion 2025-11-10 (Estimated); Study Completion 2026-01-10 (Estimated)

PRIMARY OUTCOMES:
Anxiety | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 2 days
  Self-rating scale (VAS 0-10) to rate patient anxiety, with 0 being no anxiety and 10 being extreme anxious
Symptom distress | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 2 days
  Self-rating scale (VAS 0-10) to rate symptom distress, with 0 being no distress and 10 being extreme distressed.
Relaxation | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 2 days
  Self-rating scale (VAS 0-10) to rate relaxation, with 0 being unrelaxed and 10 being very relaxed.

SECONDARY OUTCOMES:
Pulse rates | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 1 day
  The change of pulse rates during MRI scanning
Respiration rate | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 100 months
  The change of respiration rate during MRI scanning
Scanning efficiency | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 100 months
  Duration of actual scans require, duration of the whole process, and the frequency of pause due to patient in-compliance
Patient satisfaction level | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 3 days
  A 1 to 5 satisfaction scale, with 1 being strongly unsatisfied, 2 being unsatisfied, 3 being somewhere between unsatisfied and satisfied, 4 being quite satisfied. and 5 being strongly satisfied
Patient attention to music (only for the music therapy group) | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 3 days
  A 1 to 5 self-rating scale, with 1 being fully attended during the whole process, 2 being attended most time during scanning, 3 being attended sometime during scanning, 4 being unattended most time during scanning, and 5 being fully unattended

CONTACTS AND LOCATIONS:
Locations (1):
- GuangZhou Concord Cancer Center, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Undecided